CLINICAL TRIAL: NCT06929793
Title: Multiple Micronutrients Supplementation on Angiogenesis and Vasculogenesis Factors, and Fetal Biometry
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Amanda Rumondang, MD, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24081311
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-08

CONDITIONS: Angiogenesis; Fetal Weight; Pregnancy Related; Nutrient Element Deficiency; High Risk Pregnancy
Keywords: micronutrients; angiogenesis; vasculogenesis; fetal biometry
MeSH Terms: conditions — Fetal Weight

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): 1. Multiple micronutrient
  2. Calcium Carbonat 766 mg
  3. Vitamin D3 5000 IU
  4. DHA 300 mg
  Interventions: Dietary Supplement: Multiple Micronutrients
- Control (Placebo Comparator): Standard antenatal vitamins
  Interventions: Drug: Standard Antenatal Vitamin

INTERVENTIONS:
Dietary Supplement: Multiple Micronutrients — 1. Multiple micronutrient
  2. Calcium Carbonat 766 mg
  3. Vitamin D3 5000 IU
  4. DHA 300 mg
  Arms: Intervention
Drug: Standard Antenatal Vitamin — Standard Antenatal Vitamin given in Community Health Centers
  Arms: Control

SUMMARY:
Multiple micronutrients play an important role during pregnancy, since the decidualization and implantation phases. It has an impact on placentation and remodeling of blood vessels. The optimal early pregnancy conditions accompanied by great angiogenesis and vasculogenesis factors will influence fetal growth. This study aims to determine the effect of maternal multiple micronutrient supplementation on angiogenesis factors, vasculogenesis factors, and fetal biometry. It is a clustered randomized controlled trial that aims to determine the impact of maternal micronutrient supplementation on PlGF levels, sFlt-1/PlGF ratio, mean pulsatility index of uterine artery, and fetal biometry (head circumference, femur length, and estimated fetal weight percentile). The target population for the study was all pregnant women who underwent antenatal check-ups at community health centers in DKI Jakarta.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women with gestation age 8 - 14 weeks.
2. Singleton pregnancy.
3. Living in DKI Jakarta.
4. Can consume tablets or caplets.
5. Willing to only consume the vitamins used in the research
6. Willing to undergo antenatal examination at community health centers in DKI Jakarta.
7. Willing to be a research subject by signing the research consent form.

Exclusion Criteria:

1. Multiple pregnancies.
2. Pregnancy with assisted reproduction.
3. History of polycystic ovary syndrome.
4. History of chronic hypertension.
5. History of gestational diabetes mellitus.
6. Diagnosed with type 2 diabetes mellitus.
7. History of preeclampsia.
8. Recurrent miscarriage (Recurrent Pregnancy Loss).
9. Maternal medical conditions (Autoimmune; Heart Disease; Malignancy).
10. History of chronic infection.
11. Cannot consume tablets or caplets
12. Planning to move out of DKI Jakarta before and/or not giving birth in DKI Jakarta.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregant women
Enrollment: 200 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
PlGF levels | It was carried out at gestational age: 1. Trimester 1: 8-14 weeks. 2. Trimester 2: 20-26 weeks.
  Examination of angiogenesis factors in both research groups, using venous blood to measure Placental Growth Factor (PlGF) levels
sFlt-1/PlGF ratio | 20-26 weeks of gestation
  Examination of the balance of angiogenesis factors in both groups, using venous blood to measure the ratio of soluble fms-Like Tyrosine Kinase-1 to Placental Growth Factor (s-Flt-1/PlGF),
mean pulsatility index of uterine artery | 1. Trimester 1 : 8-14 weeks. 2. Trimester 2 : 20-26 weeks.
  Examination of vasculogenesis factors by measuring the mean Pulsatility Index of bilateral uterine arteries
Head circumference | 20-26 weeks of gestation
  Head circumference based on ultrasonography
Femur length | 20-26 weeks of gestation
  Femur length based on ultrasonography
Estimated fetal weight | 20-26 weeks of gestation
  Estimated fetal weight based on ultrasonography

CONTACTS AND LOCATIONS:
Locations (1):
- Maternal Fetal Medicine Division, Obstetric Gynecology Department Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided